CLINICAL TRIAL: NCT04651114
Title: Pilot Testing a New Pregnancy Decision Making Tool for Women With Physical Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Claire Z. Kalpakjian, Associate Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUM00189778; R21HD092526 (NIH)
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Results first posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-06

CONDITIONS: Disability Physical
Keywords: Medical decision making; Pregnancy, planned

STUDY DESIGN:
Intervention Model Description: A pre-post design was selected for feasibility and preliminary efficacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decision-making tool (Experimental): Women will receive the decision making tool and use for a 3 month period.
  Interventions: Behavioral: Decision-making tool

INTERVENTIONS:
Behavioral: Decision-making tool — Women will be directed to a secure website to download a copy of the decision making tool and worksheets (they can download as many copies as they wish to). The women will use the tool and worksheets at their own pace for the pilot study period.
  The decision making tool is a 23-page tool and set of 9 downloadable worksheets. The tool covers topics relevant to women with disabilities in considering or planning a pregnancy: 1) Overview of Pregnancy: 2) Knowing what is important; 3) Partners, family and important relationships; 4) Physical function and independence; 5) Health and wellbeing; 6) Caring for an infant; 7) Financial resources & insurance; 8) How to find reliable information and resources; 9) Connecting with other women with physical disabilities; 10) Dealing with reactions of others, stigma and bias, pressure; and 11) Reaching a decision.

SUMMARY:
The purpose of this project is to develop, and pilot test a decision-making tool that is tailored for women with physical disabilities to support those women in making a decision about whether or not a pregnancy is right given the participant's situation.

ELIGIBILITY:
Inclusion Criteria:

* Physical disability, defined by loss or impairment of physical function limiting one or more important life activities
* Mild, moderate or severe disability severity; severity will be assessed based on the need for assistance with daily life activities and/or personal care
* Actively planning or in the process of making a decision about whether or not to get pregnant in the near future.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Kalpakjian, PhD, MS, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Decision-making Tool: Women will receive the decision making tool and use for a 3 month period.
  Decision-making tool: Women will be directed to a secure website to download a copy of the decision making tool and worksheets (they can download as many copies as they wish to). The women will use the tool and worksheets at their own pace for the pilot study period.
  The decision making tool is a 23-page tool and set of 9 downloadable worksheets. The tool covers topics relevant to women with disabilities in considering or planning a pregnancy: 1) Overview of Pregnancy: 2) Knowing what is important; 3) Partners, family and important relationships; 4) Physical function and independence; 5) Health and wellbeing; 6) Caring for an infant; 7) Financial resources & insurance; 8) How to find reliable information and resources; 9) Connecting with other women with physical disabilities; 10) Dealing with reactions of others, stigma and bias, pressure; and 11) Reaching a decision.
Period: Overall Study
Arm/Group | Decision-making Tool
Started | 38
Completed | 30
Not Completed | 8
Not completed — Withdrawal by Subject | 8

BASELINE CHARACTERISTICS:
Arm/Group | Decision-making Tool
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 33
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38
Decisional Conflict Scale, Values Clarity sub-scale [Mean (Standard Deviation); unit: units on a scale] — The Decisional Conflict Scale is a self-report measure. Decisional conflict refers to a state of uncertainty about a course of action. For this study, this refers to uncertainty about pursuing a future pregnancy. The Values Clarity sub-scale refers to how much a respondent is clear about the values that guide their decision-making. Sub-scale items (3) are rated on 5-point Likert scales (ranging from strongly agree [5] to strongly disagree [1]) and summed for a total score range of 3 to 15. Higher scores represent greater clarity of values.
  units on a scale | 12.59 (2.3)
Decisional Conflict Scale, Support for Decision Making sub-scale [Mean (Standard Deviation); unit: units on a scale] — The Decisional Conflict Scale is a self-report measure. Decisional conflict refers to a state of uncertainty about a course of action. For this study, this refers to uncertainty about pursuing a future pregnancy. The Support for Decision Making sub-scale refers to how much support a respondent has from others about their decision-making. Sub-scale items (3) are rated on 5-point Likert scales (ranging from strongly agree [5] to strongly disagree [1]) and summed for a total score range of 3 to 15. Higher scores represent greater support for decision-making.
  units on a scale | 11.03 (3.0)
Decisional Conflict Scale, Uncertainty about the Decision sub-scale [Mean (Standard Deviation); unit: units on a scale] — The Decisional Conflict Scale is a self-report measure. Decisional conflict refers to a state of uncertainty about a course of action. For this study, this refers to uncertainty about pursuing a future pregnancy. The Uncertainty about the decision sub-scale refers to how much a respondent is uncertain about the decision. Sub-scale items (3) are rated on 5-point Likert scales (ranging from strongly agree [5] to strongly disagree [1]) and summed for a total score range of 3 to 15. Higher scores represent greater certainty about the decision.
  units on a scale | 9.37 (3.6)
Stage of Decision-Making Scale [Mean (Standard Deviation); unit: units on a scale] — The Stage of Decision Making is a single item self-report measure. The options range from "haven't begun to think about choices" to "have already made a decision and unlikely to change my mind". The instructions were modified to refer to pregnancy and excluded the first two options of not having begun to think about choices given inclusion criteria. For this study, the scale ranged from 1 (are considering the decision now) to 4 (have already made a decision and am unlikely to change my mind). A higher score reflects greater readiness to make a decision.
  units on a scale | 2.17 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Final Decisional Conflict Scale Score - Values Clarity Sub-scale
Description: The Decisional Conflict Scale is a self-report measure. Decisional conflict refers to a state of uncertainty about a course of action. For this study, this refers to uncertainty about pursuing a future pregnancy. The Values Clarity sub-scale refers to how much a respondent is clear about the values that guide their decision-making. Sub-scale items (3) are rated on 5-point Likert scales (ranging from strongly agree [5] to strongly disagree [1]) and summed for a total score range of 3 to 15. Higher scores represent greater clarity of values.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Decision-making Tool
Number analyzed (Participants) | 30
units on a scale | 13.1 (2.3)

2. Primary Outcome: Final Decisional Conflict Scale Score - Support Sub-scale
Description: The Decisional Conflict Scale is a self-report measure. Decisional conflict refers to a state of uncertainty about a course of action. For this study, this refers to uncertainty about pursuing a future pregnancy. The Support for Decision Making sub-scale refers to how much support a respondent has from others about their decision-making. Sub-scale items (3) are rated on 5-point Likert scales (ranging from strongly agree [5] to strongly disagree [1]) and summed for a total score range of 3 to 15. Higher scores represent greater support for decision-making.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Decision-making Tool
Number analyzed (Participants) | 30
units on a scale | 12.6 (2.1)

3. Primary Outcome: Final Decisional Conflict Scale Score - Uncertainty Sub-scale
Description: The Decisional Conflict Scale is a self-report measure. Decisional conflict refers to a state of uncertainty about a course of action. For this study, this refers to uncertainty about pursuing a future pregnancy. The Uncertainty about the decision sub-scale refers to how much a respondent is uncertain about the decision. Sub-scale items (3) are rated on 5-point Likert scales (ranging from strongly agree [5] to strongly disagree [1]) and summed for a total score range of 3 to 15. Higher scores represent greater certainty about the decision.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Decision-making Tool
Number analyzed (Participants) | 30
units on a scale | 11.3 (2.9)

4. Primary Outcome: Final Readiness to Make a Choice in Stage of Decision-Making Scale
Description: The Stage of Decision Making is a single item self-report measure. The options range from "haven't begun to think about choices" to "have already made a decision and unlikely to change my mind". The instructions were modified to refer to pregnancy and excluded the first two options of not having begun to think about choices given inclusion criteria. For this study, the scale ranged from 1 (are considering the decision now) to 4 (have already made a decision and am unlikely to change my mind). A higher score reflects greater readiness to make a decision.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Decision-making Tool
Number analyzed (Participants) | 30
units on a scale | 3.1 (1.0)

5. Secondary Outcome: Feasibility - Acceptability
Description: Acceptability of decision making tool is refers to whether the intervention is agreeable or satisfactory. In this study we measured this by self-report. We used 11 items that measured the presentation of information of the tool rated on Likert scales ranging from 1 (poor) to 4 (excellent) which are summed across all items. Possible scores can range from 11 to 44, with higher scores reflecting better information presentation.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Decision-making Tool
Number analyzed (Participants) | 30
units on a scale | 35.7 (6.4)

6. Secondary Outcome: Feasibility - Demand
Description: Demand refers to the likelihood of using an intervention after the study is over. For this study, it is a single item rated on Likert scales of 1 (definitely not likely) to 5 (very likely). Higher scores indicate a higher likelihood of using the tool after the study is over.
Time Frame: 12 weeks
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Decision-making Tool
Number analyzed (Participants) | 30
units on a scale | 4 (1.3)

7. Secondary Outcome: Feasibility - Ease of Use
Description: Ease of use refers to how easy an intervention is to use. In this study, we measures ease of use of the tool with a self-report, single item rated on Likert scales ranging from 1 (very hard) to 5 (very easy). A higher rating means the tool was considered easier to use.
Time Frame: 12 weeks
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Decision-making Tool
Number analyzed (Participants) | 30
units on a scale | 4.5 (1.2)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: No more than minimal risk study.
Arm/Group | Decision-making Tool
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/14/NCT04651114/Prot_SAP_000.pdf